CLINICAL TRIAL: NCT00731601
Title: Phase 4 Study of Intravenous Proton Pump Inhibitor in Patients With Peptic Ulcer Bleeding After Successful Endoscopic Therapy- a Prospective Randomized Comparative Trial
Brief Title: Intravenous Proton Pump Inhibitor for Peptic Ulcer Bleeding
Acronym: PPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Lin, Hwai-jeng, M.D. FACG, Lotung Poh-Ai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LotungPAH
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: shock; peptic ulcer bleeding; rebleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Shock | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): pantoprazole 40mg/q6h IV infusion for three days
  Interventions: Drug: pantoprazole
- 2 (Active Comparator): pantoprazole 8mg/h for three days
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole — pantoprazole 40 mg/q6h IV infusion for three days
  Other Names: pantoloc
  Arms: 1
Drug: pantoprazole — pantoprazole 8 mg/h IV infusion for three days
  Other Names: pantoloc
  Arms: 2

SUMMARY:
A large dose of PPI is effective in preventing peptic ulcer rebleeding. The investigators hypothesize that 40 mg/q6h pantoloc is equivalent to 8mg/h pantoloc in preventing rebleeding.

DETAILED DESCRIPTION:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcers and is now recommended as the first hemostatic modality for these patients.

In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies, two consensus statements and two meta-analysis. In our previous experience, we used omeprazole 160 mg /day infusion instead of 8 mg/h in these patients and obtained a good result .

The objectives of this study are to assess the outcomes of two different regimens of high dose of intravenous pantoprazole after endoscopic therapy in patients with peptic ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients were accepted for endoscopic therapy if a peptic ulcer with active bleeding, a non-bleeding visible vessel (NBVV) or an adherent blood clot at the ulcer base was observed within 24 hours of hospital admission.

Exclusion Criteria:

* If patients were pregnant
* Did not obtain initial hemostasis with endoscopic injection of epinephrine
* Did not give written informed consent
* Had bleeding tendency (platelet count < 50×109/L, serum prothrombin < 30% of normal, or were taking anticoagulants), uremia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary end point was recurrent bleeding before discharge and within 14 days. | About one year

SECONDARY OUTCOMES:
At day 14, volume of blood transfused, number of surgeries performed, and the mortality rates of the two groups are compared. | about one year

CONTACTS AND LOCATIONS:
Overall Officials: Hwai-jeng Lin, M.D., Principal Investigator — Lotung Poh-Ai Hospital
Locations (1):
- Lotung Poh-Ai hospital, Yilan, Taiwan